CLINICAL TRIAL: NCT00950586
Title: A Placebo-controlled, Single-blind, Randomised Study to Investigate the Safety, Tolerability, Pharmacokinetics and Drug Interaction of GSK1034702 After Repeat Doses in Healthy Subjects
Brief Title: Safety, Blood Levels, Drug Interaction and Effects of Repeated Doses of GSK1034702
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110792
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Cognitive Disorders
Keywords: Drug interaction; Saftey; Pharmacokinetics; Cognition
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): 14 days dosing
  Interventions: Drug: GSK1043702; Drug: Placebo
- Cohort 2 (Experimental): Single dose followed by 14 days repeat dosing
  Interventions: Drug: GSK1043702; Drug: Placebo
- Cohort 3 (Experimental): Up to 28 days repeat dosing with drug interaction
  Interventions: Drug: GSK1043702; Drug: Dextromethorphan; Drug: Placebo

INTERVENTIONS:
Drug: GSK1043702 — Oral dose in liquid or tablet formulation
Drug: Dextromethorphan — 30mg Oral dose
  Arms: Cohort 3
Drug: Placebo — To match GSK1034702

SUMMARY:
GSK1034702 is being developed for improving cognitive impairment in diseases such as Alzheimer's disease and schizophrenia. This study will be done in healthy men and women of no child beading potential to investigate repeated doses of the study medicine. The study will investigate the following questions, do repeated doses of the study medicine have any important side effects when taken by mouth? How much of the study medicine gets into the bloodstream, and how quickly does the body get rid of it? Does the study medicine affect memory, attention and problem-solving skills? What are the effects when the study medicine and dextromethorphan are taken together.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non childbearing potential
* Generally healthy
* Body mass index 19 - 29.9 kg/m2 (inclusive), body weight greater than or equal to 50 kg for males and greater than of equal to 45 kg for females
* Normal Laboratory test results

Exclusion Criteria:

* Abuse of drugs or alcohol
* Smoker or history of regular use of tobacco- or nicotine-containing products in the past 6 months
* ECG abnormality (personal or family history)
* Psychiatric disorder
* Asthma or a history of asthma
* Medical illness

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08-24 (Actual); Primary Completion 2009-12-24 (Actual); Study Completion 2009-12-24 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability endpoints consisting of: AEs; 12-lead ECG; 12 lead digital Holter and lead II telemetry; vital signs; clinical laboratory evaluations. | Up to 28 days
GSK1034702 PK parameters: Cmax; tmax; AUC(0-t) | Up to 28 days
Dextromethorphan PK parameters: Cmax; tmax; AUC(0-t). | Day -2, 1 and 14
Effects on Cognitive tests. | Up to day 28
Effects on salivary secretion | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 110792 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/110792?search=study&search_terms=110792#rs
- Available data/document: Statistical Analysis Plan: 110792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register